CLINICAL TRIAL: NCT06861972
Title: Caesarean Hysterectomy Versus Conservative Management of Placenta Accreta: A Comparative Study
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed ElHarty, Lecturer, Cairo University
Other Study IDs: MD-13-2023
Record Dates: First submitted 2025-01-14; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Obstetric Complication
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — uterine corpus in hysterectomy and areas resected out of the myometrium in focal myometrium resection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1 (Caesarean Hysterectomy group): patients with placenta accreta spectrum undergoing caesarean hysterectomy.
  Interventions: Procedure: Caesarean Hysterectomy
- 2 ( Conservative Management group): patients with placenta accreta spectrum undergoing focal myometrium resection
  Interventions: Procedure: Conservative management

INTERVENTIONS:
Procedure: Caesarean Hysterectomy — Caesarean delivery followed by hysterectomy
  Groups: 1 (Caesarean Hysterectomy group)
Procedure: Conservative management — Focal myometrium resection of the area of diseased myometrium after delivery
  Groups: 2 ( Conservative Management group)

SUMMARY:
Placenta accreta rates are rising alongside the rising rates of caesarean deliveries. This has lead to a vast number of studies negotiating the histopathological nature, risk factors and outcomes of pregnancies complicated with placenta accreta. In the study the investigators re discussing the outcome of different plans of management of placenta accreta, namely caesarean hysterectomy and focal myometrium resection.

DETAILED DESCRIPTION:
Rising rates of caesarean delivery worldwide and especially in Egypt have affected higher rates of placenta accreta spectrum disorders. The increasing prevalence of this life-threatening condition can be primarily prevented by efforts targeted at reducing primary caesarean deliveries as well as encouraging trial of labor after caesarean deliveries of carefully selected gravidas in well-equipped hospitals, capable of providing continuous electronic fetal heart rate monitoring, along with offering one to one health care based systems with the capability of performing emergency caesarean deliveries when needed. As for secondary prevention, the best surgical approach to uterine incisions in caesarean deliveries is yet to be found and universally applied. The said approach will aim at decreasing short and long term complications of uterine scarification resulting in decreased number of placenta accreta cases and possibly downgrading their difficulty, too. Having failed to prevent such occurrence, optimization of PAS management can be attempted to try and decrease implicated injuries. As previously noted, multidisciplinary systematic approach of managing placenta accreta spectrum disorders is indispensable to reduce maternal morbidity and mortality afflicted by this grave condition. The said approach begins with identification of the risk factors of PAS occurrence, calculating pretest probability of PAS and thus early suspicion and referral can be offered by the widely applicable 2nd trimester anomaly scan. After confirming the diagnosis in the 3rd trimester, birthing plans are formulated according to the gravity of the condition assessed by the patient's clinical condition, the ultrasound scan signs, together with social factors as proximity to a healthcare facility capable of offering such management alongside the maternal take on prolonged hospitalization. Decision making and choosing the place of delivery is shared between the pregnant lady, her birth companion and her following up obstetrician. Since elective management of such cases has been proven to be associated with less adjacent organ injuries and associated morbidities, late preterm delivery is usually elected after a course of antenatal corticosteroids as per local protocol.

Guidelines concerned with PAS management still consider caesarean hysterectomy as the main management of placenta accreta disorders. Owing to the high rate of associated morbidity with caesarean hysterectomy, different researchers are hunting down updated recent management approaches with less morbidity and mortality.

Our study evaluated different outcomes with conservative management of placenta accreta spectrum disorders, namely, focal myometrium resection of the adherent defective myometrium along with its overlying placenta after devascularization, as opposed to caesarean hysterectomy. Data will be observed in a total of 36 PAS patients managed in the OBGYN department, in Kasr Al-Ainy School of medicine hospital, with 18 patients undergoing the previously explained conservative management and 18 patients undergoing caesarean hysterectomy. Demographic data of both study groups, alongside operative time, adjacent organ injury estimated blood loss, need for blood transfusion, Inotropic support and ICU admission will be collected, recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy with living fetus
* Average liquor: 5-25 cm
* Gestational age ≥ 34 weeks at time of termination
* Previous lower segment cesarean section/s
* Suspected placenta accreta spectrum.

Exclusion Criteria:

* Hepatic, cardio-pulmonary or coagulation disorders

  * Hemoglobin< 9.5g/dl
  * Ruptured membranes
  * Need for emergency delivery as Antepartum hemorrhage or contractions
  * Placental abruption
  * Lower uterine segment fibroids
  * Consent withdrawal

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total number of 36 pregnant patients at or after 34 weeks diagnosed of having placenta accreta spectrum were admitted and managed in Kasr Al-Ainy School of Medicine Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
operative blood loss | 6 months
  hemoglobin deficit in mg/dl

SECONDARY OUTCOMES:
operative blood loss | 6months
  visual estimation of operative blood loss in ml
need for blood products transfusion | 6months
  no of blood products transfused in both groups in no. of units
adjacent organ injuries | 6months
  rates of urinary bladder or ureteric injuries
operative time | 6months
  operative time in minutes
ICU admission | 6months
  need for ICU admission and length of stay in days

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Collins SL, Chantraine F, Morgan TK, Jauniaux E. Abnormally adherent and invasive placenta: a spectrum disorder in need of a name. Ultrasound Obstet Gynecol. 2018 Feb;51(2):165-166. doi: 10.1002/uog.18982. No abstract available. PMID 29231264
- [Result] Nieto-Calvache AJ, Palacios-Jaraquemada JM, Osanan G, Cortes-Charry R, Aryananda RA, Bangal VB, Slaoui A, Abbas AM, Akaba GO, Joshua ZN, Vergara Galliadi LM, Nieto-Calvache AS, Sanin-Blair JE, Burgos-Luna JM; Latin American group for the study of placenta accreta spectrum. Lack of experience is a main cause of maternal death in placenta accreta spectrum patients. Acta Obstet Gynecol Scand. 2021 Aug;100(8):1445-1453. doi: 10.1111/aogs.14163. Epub 2021 May 24. PMID 33896009
- [Result] Jauniaux E, Jurkovic D. Placenta accreta: pathogenesis of a 20th century iatrogenic uterine disease. Placenta. 2012 Apr;33(4):244-51. doi: 10.1016/j.placenta.2011.11.010. Epub 2012 Jan 28. PMID 22284667
- See also: Kasr Alainy simplified uterine preserving surgery for conservative management of placenta accreta spectrum — https://pubmed.ncbi.nlm.nih.gov/37001252/
- See also: Placenta accreta spectrum: a hysterectomy can be prevented in almost 80% of cases using a resective-reconstructive technique — https://pubmed.ncbi.nlm.nih.gov/31984808/
- See also: Caesarean hysterectomy — https://pubmed.ncbi.nlm.nih.gov/23829115/